CLINICAL TRIAL: NCT04068818
Title: The Heidelberg Engineering ANTERION Imaging Agreement Study
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: B-2018-4
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Eye Abnormalities; Normal Eyes
MeSH Terms: conditions — Eye Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Eyes with normal anterior segment
  Interventions: Device: ANTERION
- Eyes with anterior segment abnormalities
  Interventions: Device: ANTERION

INTERVENTIONS:
Device: ANTERION — Biometry images will be acquired on the ANTERION and the reference device and the image quality and the identification of abnormalities will be assessed by a reading center

SUMMARY:
This is a prospective clinical study that will be conducted at one clinical site located in the United States to assess image quality of acquired biometry images of the eye

DETAILED DESCRIPTION:
The conducted study is a non-interventional study for an imaging device used in the aid of ophthalmology diagnosis. Because the study is not interventional, the study is not an Applicable Clinical Trial per Clinicaltrials.gov definition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 years or older
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions
3. Able to fixate
4. With eye pathology status for each of the two eye populations. A. Eye with normal anterior segment

B. Eyes with anterior segment abnormalities identified with the slit lamp exam including but not limited to:

* glaucoma surgeries: trabeculectomy, laser peripheral iridotomy and drainage devices
* corneal surgeries: corneal inlays and corneal transplants
* pterygium and corneal scar

Exclusion Criteria:

1. Subjects which were enrolled in the B-2018-1 Study
2. Physical inability to be properly positioned at the study devices or eye exam equipment
3. Contact lenses worn during imaging

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A: normal eyes B: eyes with anterior segment abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Image quality | 30 days
  Comparison of the B-Scan image quality between the ANTERION and the reference device
Agreement in identification of abnormality | 30 days
  Agreement in identification of abnormality from OCT B-Scan images between ANTERION and the reference device

SECONDARY OUTCOMES:
Adverse Events | 1 day
  Evaluate any adverse events found during the clinical study

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Dul, Principal Investigator — State University of New York College of Optometry
Locations (1):
- State University of New York College of Optometry, New York, New York, United States